CLINICAL TRIAL: NCT03154840
Title: A Randomized, Open Label, Single Subcutaneous Dose 6x3 Crossover Study to Investigate the Relative Bioavailability Among Different Eutropin Formulations in Healthy Male Volunteers
Brief Title: Relative Bioavailability Among Different Eutropin Formulations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: LG-HGCL009
Record Dates: First submitted 2017-04-25; First posted 2017-05-16 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Relative Bioavailability

STUDY DESIGN:
Intervention Model Description: 6x3 Crossover Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eutropin 4IU (Experimental)
  Interventions: Drug: Eutropin 4IU, Eutropin AQ 12IU, Eutropin Pen 36IU
- Eutropin AQ 12IU (Experimental)
  Interventions: Drug: Eutropin 4IU, Eutropin AQ 12IU, Eutropin Pen 36IU
- Eutropin Pen 36IU (Experimental)
  Interventions: Drug: Eutropin 4IU, Eutropin AQ 12IU, Eutropin Pen 36IU

INTERVENTIONS:
Drug: Eutropin 4IU, Eutropin AQ 12IU, Eutropin Pen 36IU — Investigate the Relative Bioavailability among Different Eutropin Formulations

SUMMARY:
1. Compares and evaluates the relative bioavailability of single-dose subcutaneous administration of each of the Eutropin formulations to healthy male volunteers.
2. Ensure safety and tolerability of single, subcutaneous administration of Eutropin formulations to healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy male who is at least 19 years old but under 40 years of age at screening visit
2. Those who weigh more than 50 kg at screening visit and whose body mass index (BMI) is greater than 19 kg / m2 but less than 28 kg / m2
3. The result of the vital signs in the screening period.
4. A person who is judged to be clinically insignificant in terms of physical or mental condition when the examinee medically judges the screening period physical examination
5. Those who are not clinically significant when the examiner has medically judged the results of examination other than the items described in 17) and 18) of the exclusion criterion in the diagnosis laboratory test results in the screening period
6. A person who consents to use a combination of effective contraceptive methods or medically appropriate contraceptive methods from the first administration of the clinical trial drug to the fourth administration (28 days) after the last administration of the drug for clinical trial and not to provide sperm
7. Those who voluntarily decide to participate in clinical trials and observe the test subjects' precautions and agree in writing

Exclusion Criteria:

1. Those who with a history or history of diabetes
2. Those who with a history or history of malignancy
3. Those who with a history or history of musculoskeletal disorders (including epiphyseal closure, scoliosis, etc.)
4. Those who with history or history of endocrine system (including hypothyroidism, panhypopituitarism, etc.)
5. Those who have a history of skin disease, including psoriasis and contact dermatitis, or who can not exclude the possibility of skin disease under the judgment of the examiner on physical examination conducted at the screening visit.
6. Exclusion Criteria In addition to items 1) to 5), there are other clinically significant history or history of liver, kidney, digestive system, respiratory system, neuropsychiatry, blood /
7. Persons with a history of somatropin and octreotide acetate or hypersensitivity reactions to cresol, glycerol or other drugs (non-steroidal anti-inflammatory drugs, antibiotics, etc.)
8. Those who have participated in other clinical trials or bioequivalence tests within 90 days of the screening visit date
9. Within 60 days before screening visit Those who have received blood (blood, whole blood, etc.) or blood transfusions
10. Those who ingest herbal medicines or health functional foods within 14 days before the screening visit or those who are expected to affect the clinical trial within 7 days
11. Within 14 days prior to screening visit, special medicines that may affect the clinical trial, or those who use general medicines within 7 days
12. Screening Within 30 days prior to the visiting date Alcohol Abuse (alcohol-containing beverage> 21 units / week)
13. Over 30 days before screening visit Overcame smoker (cigarette> 10 cigarettes / day)
14. Within 7 days of screening visit Caffeine-containing foods Excessive intake (caffeinated foods> 3 times / week)
15. Screening Within 7 days prior to the visit Date of intake of food containing xanthine
16. As a result of urine nicotine test or urine drug screening test during the screening period
17. Screening period serum test (hepatitis B test, human immunodeficiency virus (HIV) test, hepatitis C test, syphilis test) Result positive
18. Diagnosis of Screening Period In the case of a laboratory test, one or more of the following findings

    * Fasting glucose> 110 mg / dL
    * TSH Reference Range Above upper limit or below lower limit
    * IGF-1 and IGFBP-3 according to the age of the test subjects. Reference range Above upper limit or below lower limit
    * Vitamin B12 Reference range above or below the upper limit
    * Insulin reference range above or below the upper limit
    * More than twice the AST or ALT or Alkaline Phosphatase (ALP) reference range upper limit
    * More than 1.5 times the upper limit of the bilirubin total reference range
19. A 12-electrode electrocardiogram in the screening period revealed a QTc> 450 ms or clinically significant abnormalities
20. Those who are judged to be inadequate to perform the clinical trial when the examiners judge them for other reasons

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-11-30 (Estimated)

PRIMARY OUTCOMES:
AUClast of somatropin | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacokinetic assessment

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of somatropin | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacokinetic assessment
Area under the plasma concentration versus time curve (AUCinf) of somatropin | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacokinetic assessment
Time at which the Cmax is observed (Tmax) of somatropin | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacokinetic assessment
Elimination half-life time (t1/2β) of somatropin | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacokinetic assessment
IGF-1 | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacodynamic assessment
IGF-BP3 | Total three period at weekly intervals (Week 1, Week2, Week3)
  Pharmacodynamic assessment
Monitoring of adverse reactions | Week -4(Screening), Week 1, Week 2, Week 3, Week 5
  Clinical significance is assessed by reviewing the general findings of individual subjects individually, and when there is a specific or tendency, analysis is conducted
Physical examination | Week -4(Screening), Week 1, Week 2, Week 3, Week 5
  Weight, Height
Vital Signs | Week -4(Screening), Week 1, Week 2, Week 3, Week 5
  Left-sided blood pressure (systolic / diastolic), pulse rate, tympanic temperature
Electrocardiogram | Week -4(Screening), Week 1, Week 2, Week 3, Week 5
  Ventricular rate, PR interval, QRS, QT/QTc
Laboratory test | Week -4(Screening), Week 1, Week 2, Week 3, Week 5
  General blood test, general chemical test, clinical chemistry urinalysis, pancreas test
Injection site reaction and Pain scale evaluation | Week 1, Week 2, Week 3
  Ask the NRS about the degree of pain and evaluate it as 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Asan Medical Center, Seoul, South Korea